CLINICAL TRIAL: NCT06650072
Title: Palatal vs Tuberosity Micro-connective Tissue Grafts for the Treatment of Multiple Adjacent Gingival Recession Defects: a Multi-center Controlled Randomized Clinical Trial
Brief Title: Effectiveness of Tuberosity Micro Connective Tissue Graft for Treatment of Multiple Adjacent Gingival Recession Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCarcuac-tuberosity microCTG
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palatal Micro Connective Tissue Graft (Active Comparator): A mucogingival surgery where a connective tissue graft harvested from the palate is divided in multiple micro connective tissue grafts and placed on a recipient site prepared for modified coronally advanced tunnel and sutured to cover multiple adjacent gingival recession defects.
  Interventions: Procedure: modified coronally advanced tunnel technique combined with multiple palatal micro connective tissue grafts
- Tuberosity Micro Connective Tissue Graft (Experimental): A mucogingival surgery where a connective tissue graft harvested from the maxillary tuberosity is divided in multiple micro connective tissue grafts and placed on a recipient site prepared for modified coronally advanced tunnel and sutured to cover multiple adjacent gingival recession defects.
  Interventions: Procedure: modified coronally advanced tunnel technique combined with multiple tuberosity micro connective tissue grafts

INTERVENTIONS:
Procedure: modified coronally advanced tunnel technique combined with multiple palatal micro connective tissue grafts — The connective tissue graft will be harvested from the palate.
  Arms: Palatal Micro Connective Tissue Graft
Procedure: modified coronally advanced tunnel technique combined with multiple tuberosity micro connective tissue grafts — The connective tissue graft will be harvested from the maxillary tuberosity.
  Arms: Tuberosity Micro Connective Tissue Graft

SUMMARY:
The objective of this project is to compare post-operative pain associated with palatal and tuberosity donor sites for micro-CTG, and to evaluate the outcomes in both the donor and recipient sites.

DETAILED DESCRIPTION:
A variety of surgical methods have been reported to reestablish root coverage, including tunneling techniques and coronally and laterally advanced flaps. As thin gingival tissue is one of the predisposing factors for GRD, the adjuvant use of subepithelial connective tissue grafts (CTGs) is often considered. CTGs are thought to contribute to phenotype modification and stability of treatment outcomes and studies have indicated favorable esthetic results and high degrees of root coverage. CTGs are preferably harvested either from the lateral superficial part of the palate or from the tuberosity, due to the high amount of lamina propria and minimal submucosal tissue (adipose and glandular tissue).

When multiple adjacent teeth exhibit GRDs, the preferred surgical approach should offer the greatest possible root coverage, while limiting drawbacks (i.e., patient morbidity, esthetic problems). Thus, one of the challenges related to coverage of multiple GRDs is the scarcity of donor tissue. Modification of the harvested CTG into multiple "micro-CTG" has been proposed for the treatment of multiple adjacent GRDs (MAGRD) in order to reduce the amount of CTG to be harvested. Soft-tissue grafts from the tuberosity are increasingly gaining popularity not only because they are easier to harvest, are denser in connective tissue fibers but also because harvesting from the tuberosity presents minimal risk of intra- or post-operative complications, resulting in reduced patient morbidity. However CTG from maxillary tuberosity have been reported to induce a hyperplastic response in some patients.

The objective of this study will be to compare palatal versus tuberosity micro-CTG on postoperative pain, oral health-related quality of life (OHRQoL), degree of root coverage and esthetic outcomes.

The investigators hypothesise that no statistically significant differences will be observed in terms of %root coverage and patient satisfaction at 12 months (non-inferiority). Subjects in the test group (micro-CTG) will report significantly lower morbidity at 1 and 2 weeks post-surgery when compared to controls (superiority).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* systemically healthy,
* presenting adjacent RT1/RT2 recessions, on both sides of the anterior maxilla, with an apico-coronal extension (i.e. recession depth) > 2mm combined with thick phenotype and deep root concavity.

Exclusion Criteria:

* pregnancy or lactation,
* heavy tobacco smoking (>15 cigarettes/day),
* uncontrolled medical conditions and intake of medication that can affect gingival conditions.
* uncorrected trauma from toothbrushing,
* severe tooth malposition,
* history of root coverage procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean mid-facial recession coverage (mRC) | up to 1 year
  Percentage of the exposed tooth root covered after surgical intervention

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | up to 1 year
  Frequency of complete root coverage
Changes of Keratinized Tissue Width (KTW) | up to 1 year
  Measured as the distance from the muco-gingival-junction to the gingival margin
Changes of Gingival Thickness (GT) | up to 1 year
  Measured 3 mm apically from the free gingival margin at the mid-buccal aspect of the tooth
Patient Morbidity/Discomfort | up to 2 weeks
  Measured using an oral health-related quality of life questionnaire (OHRQoL)
Patient Satisfaction | up to 1 year
  Measured with Visual Analogue Scale (VAS), which consists of a 10cm line, with two end points representing 0 ('not satisfied') and 10 ('satisfied as much as it could possibly be')

CONTACTS AND LOCATIONS:
Overall Officials: Jan Derks, DDS, PhD, Study Chair — Goteborg University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Result] Sanz-Martin I, Rojo E, Maldonado E, Stroppa G, Nart J, Sanz M. Structural and histological differences between connective tissue grafts harvested from the lateral palatal mucosa or from the tuberosity area. Clin Oral Investig. 2019 Feb;23(2):957-964. doi: 10.1007/s00784-018-2516-9. Epub 2018 Jun 18. PMID 29915931
- [Result] Dellavia C, Ricci G, Pettinari L, Allievi C, Grizzi F, Gagliano N. Human palatal and tuberosity mucosa as donor sites for ridge augmentation. Int J Periodontics Restorative Dent. 2014 Mar-Apr;34(2):179-86. doi: 10.11607/prd.1929. PMID 24600654
- [Result] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093